CLINICAL TRIAL: NCT03430154
Title: Awareness, Care, and Treatment In Obesity Management of Patients With Hemophilia (ACTION) to Inform Hemophilia Obesity Patient Empowerment (HOPE)
Acronym: ACTION to HOPE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: HAEM-4414; U1111-1199-8271 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-01-16; First posted 2018-02-12 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Haemophilia A, Haemophilia B, Obesity
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Adults with hemophilia and obesity/overweight: Adults (any gender) aged ≥18 years with hemophilia (any severity, with or without inhibitors) self-identified with obesity or overweight
  Interventions: Other: No treatment given
- Caregivers identified with obesity/overweight: Caregivers of children (any gender) currently aged <18 years with hemophilia (any severity, with or without inhibitors) caregiver-identified with obesity or overweight
  Interventions: Other: No treatment given
- Spouses or partners self-identified with obesity/overweight: Spouses or partners of adults (any gender) aged ≥18 years with hemophilia (any severity, with or without inhibitors) self-identified with obesity or overweight
  Interventions: Other: No treatment given
- Healthcare profs. managing hemophilia and obesity/overweight: Healthcare professional (pediatric or adult hematologist, nurse, nurse practitioner, physician assistant, physical therapist, social worker) actively working in a federally designated hemophilia-treatment center for at least 3 years and with experience managing patients with hemophilia and obesity or overweight.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
An online web-based cross-sectional survey in which participants will complete a distinct questionnaire for patients with hemophilia and obesity (PwHO) and/or their carers/spouses/partners, or a distinct questionnaire for healthcare professionals. Each questionnaire consists of more than 100 items including pre-coded (multiple choice) closed-ended questions, yes/no questions and rating scales. It is estimated that this one-off survey will take approximately 45-60 minutes to complete.

As a cross-sectional study, there will be no treatment of patients.

ELIGIBILITY:
Inclusion Criteria:

* Meeting one of the following criteria: a) Adults (any gender) aged equal to or more than 18 years with hemophilia (any severity, with or without inhibitors) self-identified with obesity or overweight, - OR - Caregivers of children (any gender) currently aged less than18 years with hemophilia (any severity, with or without inhibitors) caregiver-identified with obesity or overweight, - OR - Spouses or partners of adults (any gender) aged equal to or more than 18 years with hemophilia (any severity, with or without inhibitors) self-identified with obesity or overweight - OR - Healthcare professional (pediatric or adult hematologist, nurse, nurse practitioner, physician assistant, physical therapist, social worker) actively working in a federally designated hemophilia-treatment center for at least 3 years and with experience managing patients with hemophilia and obesity or overweight.
* Participants must have access to the internet, either at home or at a location convenient to them
* Provision of informed consent before the start of any survey-related activities.

Exclusion Criteria:

* Inability to understand and comply with written instructions in English
* Previous completion of this study with receipt of compensation
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with hemophilia and obesity/overweight, their caregivers/spouses/partners, and their healthcare providers (HCPs)
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-04-29 (Actual); Study Completion 2018-04-29 (Actual)

PRIMARY OUTCOMES:
Prevalence of obesity awareness and perceptions | Start of interviews day 1 until end of data collection day 90
  Data is collected via online questionnaires
Prevalence of attitudes on obesity | Start of interviews day 1 until end of data collection day 90
  Data is collected via online questionnaires
Prevalence of weight loss support structure | Start of interviews day 1 until end of data collection day 90
  Data is collected via online questionnaires
Prevalence of interactions between patients and HCPs around obesity/overweight | Start of interviews day 1 until end of data collection day 90
  Data is collected via online questionnaires
Prevalence of awareness about weight loss solutions | Start of interviews day 1 until end of data collection day 90
  Data is collected via online questionnaires
Characteristics of obesity awareness and perceptions | Start of interviews day 1 until end of data collection day 90
  Data is collected via online questionnaires
Characteristics of attitudes on obesity | Start of interviews day 1 until end of data collection day 90
  Data is collected via online questionnaires
Characteristics of weight loss support structure | Start of interviews day 1 until end of data collection day 90
  Data is collected via online questionnaires
Characteristics of interactions between patients and HCPs around obesity/overweight | Start of interviews day 1 until end of data collection day 90
  Data is collected via online questionnaires
Characteristics of awareness about weight loss solutions | Start of interviews day 1 until end of data collection day 90
  Data is collected via online questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure' (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Plainsboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/website/content/how-to-access-clinical-trial-datasets.aspx